CLINICAL TRIAL: NCT01360177
Title: Radioactive Iodide (131I) Treatment of 124I PET/CT Detected Breast Cancers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRSMTS0012; SU-07292008-1271 (Other: Stanford University); 14941 (Other: Stanford IRB)
Record Dates: First submitted 2011-04-18; First posted 2011-05-25 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radioactive Iodide and PET/CT (Experimental)
  Interventions: Procedure: 124 PET/CT imaging; Drug: Na134I; Drug: Tri-iodothyronine

INTERVENTIONS:
Procedure: 124 PET/CT imaging — Standard of Care
  Other Names: Positron emission tomography - computed tomography
Drug: Na134I — 25 to 150 mCi
  Other Names: GE Healthcare
Drug: Tri-iodothyronine — 75 ug/8hr x 4 weeks; oral
  Other Names: T3
Drug: Tri-iodothyronine — 20 mg/day x 2
  Other Names: T3

SUMMARY:
This is a treatment protocol designed to accompany the ongoing institutional 124I PET/CT pilot imaging study for patients with invasive breast cancer. Women whose tumors express NIS [Na+I- symporter, sodium iodide symporter] and demonstrate radioiodide uptake on 124I PET/CT scans will be eligible for 131I treatment if, (1) tumor dosimetry calculations yield a cumulative radiation dose of at least 30Gy in target tumor, (2) estimated cumulative thyroid irradiation is less than 500 cGy and, (3) the therapeutic dose of 131I is in the range of 25 to 100 mCi.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable locally advanced or metastatic breast cancer who completed 124I PET/CT imaging study.
* Patients who are 18 years of age or older.
* Patients must have a life expectancy of at least 3 months.
* I 124 dosimetry completed with thyroid dose to 500 cGy or less and tumor dose of 2500 cGy or more.
* I131 therapeutic dose calculated from dosimetry. Dose must be in a range of 25 to 150 mCi.
* Patients with Eastern Cooperative Oncology Group (ECOG) Performance Status 0-3 will be eligible.
* Use of concurrent systemic therapy (hormonal or cytotoxic) if associated with stable disease for at least three months prior to treatment.
* Women with locally advanced breast cancer and simultaneous metastases, even if surgery to eradicate local disease has taken place.
* Thyroid stimulating hormone (TSH) must be < 0.4 uIU/mL.
* White blood cell count >= 1,500 and platelet count >= 40,000
* Women receiving thyroid hormone supplements and methimazole.
* Ability to understand and the willingness to sign a written informed consent document.
* Premenopausal women must use contraception while receiving this treatment and during follow-up period of 42 days.

Exclusion Criteria:

* Stage 0-II breast cancer.
* Pregnant or nursing women.
* Not able to sign informed consent.
* Untreated psychiatric disorder.
* Women who have not had I124 PET/CT scan and dosimetry calculations.
* Radioiodide uptake in non-target organs or bone marrow does not exceed 25 cGy by pre-treatment dosimetry.
* Received chemotherapy less than 4 weeks before.
* History of thyroid cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Target lesion size will be assessed clinically or radiologically in two directions . RECIST (Response Evaluation Criteria In Solid Tumors) will be implemented to determine response | 6 WEEKS POST-TREATMENT
  * cCR (complete clinical response) = disappearance of all tumor
  * cPR (clinical partial response) = >=30% decrease sum of longest target lesion diameters
  * cPD (progressive disease) = >=20% increase sum of longest target lesion diameters.
  * cSD (stable disease) = small changes that do not meet these criteria

SECONDARY OUTCOMES:
Non target lesion size will be assessed clinically or radiologically in two directions . RECIST (Response Evaluation Criteria In Solid Tumors) will be implemented to determine response | EVALUATED AT 6 WEEKS
  * Complete Response (CR): Disappearance of all non-target lesions
  * Incomplete Response/Stable Disease (SD): Persistence of one or more non-target lesions(s)
  * Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions

CONTACTS AND LOCATIONS:
Overall Officials: Irene L. Wapnir, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States